CLINICAL TRIAL: NCT05162222
Title: An Open-label, Randomized, 2-Period Crossover Study to Evaluate the Effect of Co-administration of Itraconazole or Diltiazem on the Single-dose Pharmacokinetics of Danicamtiv in Healthy Participants
Brief Title: A Study to Evaluate the Effect of Co-administration of Itraconazole or Diltiazem on the Single-dose of Danicamtiv in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV028-008
Record Dates: First submitted 2021-12-09; First posted 2021-12-17 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-07

CONDITIONS: Healthy Participants
Keywords: Danicamtiv; Itraconazole; Diltiazem; BMS-986434; CYP3A4
MeSH Terms: interventions — Itraconazole; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Danicamtiv, followed by itraconazole + danicamtiv (Experimental)
  Interventions: Drug: Danicamtiv; Drug: Itraconazole
- Danicamtiv, followed by diltiazem + danicamtiv (Experimental)
  Interventions: Drug: Danicamtiv; Drug: Diltiazem

INTERVENTIONS:
Drug: Danicamtiv — Specified dose on specified days
Drug: Itraconazole — Specified dose on specified days
  Arms: Danicamtiv, followed by itraconazole + danicamtiv
Drug: Diltiazem — Specified dose on specified days
  Arms: Danicamtiv, followed by diltiazem + danicamtiv

SUMMARY:
The purpose of this study is to evaluate the effects of co-administration of itraconazole or diltiazem on the single-dose pharmacokinetics of danicamtiv in healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Body mass index between 18 and 30 kg/m^2, inclusive, at the Screening Visit
* Normal ECG at the Screening Visit
* Normal renal function at Screening

Exclusion Criteria:

* History of ventricular arrhythmias
* History of heart disease or conduction disorders
* History of dizziness and/or recurrent headaches (ie, daily headaches lasting for a 1-week duration in the last month prior to study intervention administration)

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 17 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time ((AUC(INF)) | Up to 17 days
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration ((AUC(0-T)) | Up to 17 days

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Up to 17 days
Concentration at 24 hours (C24) | Up to 17 days
Apparent terminal plasma half-life (T-HALF) | Up to 17 days
Incidence of adverse events (AEs) | Up to 28 days
Incidence of serious adverse events (SAEs) | Up to 28 days
Incidence of participants with vital sign abnormalities | Up to 17 days
Incidence of participants with electrocardiogram (ECG) abnormalities | Up to 17 days
Incidence of participants with physical exam abnormalities | Up to 17 days
Incidence of participants with clinical laboratory abnormalities | Up to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit - Dallas, Dallas, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm